CLINICAL TRIAL: NCT03782051
Title: Combined Phacoemulsification and Viscocanalostomy With Ologen Implant Versus Combined Phacoemulsification and Viscocanalostomy
Brief Title: Combined Viscocanalostomy, Phacoemulsification, OIogen Implant in Open Angle Glaucoma
Acronym: Visco-ologen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed moamen, princibal investigator, lecturer of ophthalmology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1102108
Record Dates: First submitted 2018-12-16; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Viscocanalostomy; Ologen; glaucoma; phacoemulsification
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — collagen-glycosaminoglycan copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phacovisco group (Active Comparator): group had combined phacoemulsification and viscocanalostomy
  Interventions: Procedure: combined phacoemulsification and viscocanalostomy
- OloPhacovisco group (Active Comparator): group had combined phacoemulsification and viscocanalostomy and Ologen
  Interventions: Procedure: combined phacoemulsification and viscocanalostomy and ologen

INTERVENTIONS:
Procedure: combined phacoemulsification and viscocanalostomy — phacoemulsification with viscocanalostomy
  Other Names: phaco-visco-canalostomy
  Arms: Phacovisco group
Procedure: combined phacoemulsification and viscocanalostomy and ologen — phacoemulsification with viscocanalostomy with ologen
  Other Names: phaco-visco-canalostomy with ologen implant
  Arms: OloPhacovisco group

SUMMARY:
This prospective, interventional, randomized clinical study was done at Alpha Vision Center, Zagazig, Egypt. Patients with coexisting cataract and glaucoma were randomized to receive either phaco-viscocanalostomy (Phacovisco group) or phaco-viscocanalostomy with Ologen® implant (OloPhacovisco group) . Follow-up period was 2 years. Nd:YAG laser goniopuncture was done in cases where the intraocular pressure (IOP) was elevated above 21 mmHg after discontinuation of corticosteroid eye drops at any follow-up visit.

Our hypothesis is that using Ologen® implant as a spacer in the subscleral reservoir in phaco-viscocanalostomy reduces fibrosis and increase the success rate of this operation

DETAILED DESCRIPTION:
Background: To study the efficacy of the biodegradable collagen implant Ologen® as an adjuvant in phaco-viscocanalostomy in patients with coexisting cataract and primary open angle glaucoma.

Methods: This prospective, interventional, randomized clinical study was done at Alpha Vision Center, Zagazig, Egypt. Patients with coexisting cataract and glaucoma were randomized to receive either phaco-viscocanalostomy (Phacovisco group) or phaco-viscocanalostomy with Ologen® implant (OloPhacovisco group). Follow-up period was 2 years. Nd:YAG laser goniopuncture was done in cases where the intraocular pressure (IOP) was elevated above 21 mmHg after discontinuation of corticosteroid eye drops at any follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* the presence of significant cataract interfering with vision (visual acuity ≤ 0.5) in the presence POAG.
* if cataract was associated with uncontrolled glaucoma, (IOP > 21 mmHg despite maximally tolerated medical therapy)
* if the IOP was ≤ 21 mmHg with use of at least two antiglaucoma drugs with medication intolerance
* poor patient compliance
* patients could not attend medical supervision
* patients had visual field deterioration.

Exclusion Criteria:

* closed-angle glaucoma
* other types of open angle glaucoma (OAG), e.g. pigmentary glaucoma, inflammatory glaucoma or neovascular glaucoma,
* previous ocular trauma or surgery
* lens subluxation
* any eye diseases affecting the vision, e.g. anterior uveitis
* if there was a large perforation of the Descemet's membrane with iris prolapse during surgery (cases with microperforation, which is defined as small perforation with no associated iris prolapse, occurring during surgery were not excluded) intraoperative complications that might affect the IOP, e.g. vitreous loss.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-01-14 (Actual); Study Completion 2018-01-14 (Actual)

PRIMARY OUTCOMES:
the intraocular pressure | 2 years
  measured by mmHg using Goldman applanatin tonometry

SECONDARY OUTCOMES:
surgical complications | 2 years
  number of surgical complications encountered
the use and results of Nd:YAG laser goniopuncture | 2 years
  number of cases needed goniopuncture
visual acuity results | 2 years
  visual acuity measured by decimal system

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AM Gad, MD, Principal Investigator — Zagazig University
Locations (1):
- Alpha vision center, Zagazig, Al Sharkeya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cillino S, Di Pace F, Cillino G, Casuccio A. Biodegradable collagen matrix implant vs mitomycin-C as an adjuvant in trabeculectomy: a 24-month, randomized clinical trial. Eye (Lond). 2011 Dec;25(12):1598-606. doi: 10.1038/eye.2011.219. Epub 2011 Sep 16. PMID 21921953
- [Background] Narayanaswamy A, Perera SA, Htoon HM, Hoh ST, Seah SK, Wong TT, Aung T. Efficacy and safety of collagen matrix implants in phacotrabeculectomy and comparison with mitomycin C augmented phacotrabeculectomy at 1 year. Clin Exp Ophthalmol. 2013 Aug;41(6):552-60. doi: 10.1111/ceo.12058. PMID 23279607
- [Background] Johnson MS, Sarkisian SR Jr. Using a collagen matrix implant (Ologen) versus mitomycin-C as a wound healing modulator in trabeculectomy with the Ex-PRESS mini glaucoma device: a 12-month retrospective review. J Glaucoma. 2014 Dec;23(9):649-52. doi: 10.1097/IJG.0000000000000018. PMID 24240882
- [Background] Hondur A, Onol M, Hasanreisoglu B. Nonpenetrating glaucoma surgery: meta-analysis of recent results. J Glaucoma. 2008 Mar;17(2):139-46. doi: 10.1097/IJG.0b013e31814b98f7. PMID 18344761
- [Background] Shaarawy T, Mermoud A. Deep sclerectomy in one eye vs deep sclerectomy with collagen implant in the contralateral eye of the same patient: long-term follow-up. Eye (Lond). 2005 Mar;19(3):298-302. doi: 10.1038/sj.eye.6701469. PMID 15258610
- [Derived] Gad AAM, Abdulhalim BH, Lotfy A, Abdelrahman AM, Ahmed AS. Combined phacoemulsification and viscocanalostomy with Ologen implant versus combined phacoemulsification and viscocanalostomy. BMC Ophthalmol. 2019 Feb 6;19(1):45. doi: 10.1186/s12886-019-1049-6. PMID 30727982

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03782051/Prot_SAP_000.pdf